CLINICAL TRIAL: NCT01581424
Title: Natural History and Structural Functional Relationships in Fabry Renal Disease Natural History, Structural Functional Relationships and Determinants of Renal Structural Responses (Changes) With Enzyme Replacement Therapy in Fabry Disease
Brief Title: Natural History and Structural Functional Relationships in Fabry Renal Disease Treatment Outcomes(Changes)in Fabry Renal Disease Study
Acronym: LDN6702
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Washington University School of Medicine (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 100349; U54NS065768 (NIH)
Record Dates: First submitted 2012-01-17; First posted 2012-04-20 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Fabry Disease
Keywords: Fabry disease; kidney function; kidney structure morphometry; Fabry kidney disease; Podocytes
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma samples as well as urine samples from an overnight collection.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will perform a study with two major components. The first is a natural history study of untreated Fabry patients. This study component will detail kidney microscopic structural changes in Fabry patients before starting enzyme replacement therapy and will correlate these changes with kidney function, including glomerular filtration rate and urinary albumin excretion rate. The investigators will perform studies on samples obtained at baseline, or before enzyme replacement therapy is initiated. The goal of our study is to find kidney microscopic changes in the biopsies that are associated with kidney disfunction. Our hypotheses for this study are:

1. Much of the natural history of Fabry renal structural changes will occur without detectable renal functional alterations.
2. Structural changes associated with the initial onset of proteinuria and those associated with the subsequent progressive loss of filtration function will differ and will be best described by non-linear models.
3. There will be sufficient precision of Fabry renal structural-functional relationships to support renal structure as an acceptable clinical trial surrogate endpoint for later renal functional deterioration.

The second component examines the effects of age and gender at start of enzyme replacement therapy (ERT), as well as dosage levels of ERT on the renal cellular clearance of GL3 from Fabry patients by comparing baseline to follow-up kidney biopsies performed 5, 11, and 60 months later, with all comparisons matched for ERT treatment duration. Our hypotheses for this component of the study are as follows:

1. Enzyme Replacement Therapy(ERT) instituted at younger ages is more effective in reducing podocytes(PC),distal tubular cells(DTC),and arterial smooth muscle cells (ASMC)GL-3 than in older Fabry patients.
2. Earlier institution of ERT will stabilize PC numbers while later ERT institution, especially in proteinuric adults, may not prevent progressive decline in PC numbers and associated glomerular sclerosis, tubulointerstitial injury, and GFR loss.
3. Whereas lower ERT dose may effectively clear GL-3 from endothelial and mesangial cells, it will be less effective in clearing GL-3 from PC and also from DTC and ASMC.
4. Affected cells will be cleared of GL-3 equivalently in females and males.

DETAILED DESCRIPTION:
Fabry disease is a rare genetic disease with deficient activity of enzyme alpha-galactosidase A. Deficient activity of this enzyme leads to the accumulation of lipid-derived inclusions in different organs including kidney, heart and vessels. These inclusions can be found in the kidney even before birth. The earliest known clinical manifestation of Fabry kidney disease is the appearance of excess protein in the urine, which usually occurs in the second decade of life. However, our studies, as well as those of other investigators show evidence that kidney injury starts much earlier. Once excess protein is found in the urine, kidney function deterioration becomes progressive, and most Fabry patients require kidney transplantation or hemodialysis in the third to fifth decade of life. The lesion or composite of lesions responsible for functional deterioration of the kidney in Fabry disease are not well known. Their delineation using quantitative, unbiased, morphometric methods will help to understand this disease, and to develop surrogate structural outcomes for early intervention trials. Enzyme replacement therapy may stabilize kidney function. However, its long-term effect on kidney survival is not known. Moreover, there is no early known predictor of kidney dysfunction to adjust and evaluate effectiveness of enzyme replacement therapy. Our studies of renal GL-3 clearance comparing pre-and post-ERT renal biopsies using the above methods will allow us to determine whether age at institution of treatment and ERT dose affect ERT induced GL-3 cellular clearance, especially from those cells where ERT is less effective, i.e., podocytes, vascular smooth muscle cells and distal tubular cells. Finally, it is our hypothesis that mosaicism in Fabry disease females is such that cells such as podocytes are either affected or normal and that ERT clearance in the affected podocytes in females will, as in males, be dependant on age of institution of treatment and ERT dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Fabry disease who have/have not received enzyme replacement therapy where a clinical decision has been made to obtain a kidney biopsy, a GFR, and urinary albumin studies or where patients have previously completed clinical trials which included measures of renal function and renal biopsies.

Exclusion Criteria:

* Patients with serum creatinine more than 2.5 mg/dL or known to have a renal disease other than Fabry.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50-60 male and female adults and children with Fabry disease who either have or have not been initiated on enzyme replacement therapy, and whose physicians have determined that a kidney biopsy and renal functional studies are clinically indicated before initiation of enzyme replacement therapy and as follow-up for this therapy or who have completed clinical trials of ERT, have baseline or baseline and and follow biopsies, and have consented to allow their tissues to be examined for research purposes. We are expecting to recruit patients from many different centers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Natural History and Determinants of Renal Structural Responses (Changes) to Enzyme Replacement Therapy in Fabry Disease | Natural history component, cross sectional; ERT component, 5, 11, and 60 months
  Renal function measurements for the cross sectional natural history component will be urine protein excretion and measured/estimated GFR. Renal biopsies will provide estimates of the amount of GL-3 in various kidney structures. We will determine which structural parameter or composite of structural parameters is most closely associated with kidney function. For renal structural responses (changes) with ERT the primary outcome will the magnitude of reduction in podocyte GL-3 per glomerulus after (a)5 months, (b) 11 months, and (c) 60 months of ERT.

SECONDARY OUTCOMES:
Natural History and Determinants of Renal Structural Responses (Changes) to Enzyme Replacement Therapy in Fabry Disease | Baseline, 5, 11 and 60 months
  The secondary endpoint for the determinants of renal structural responses to ERT will be GL-3 reduction from baseline to 5, 11 and 60 months in a composite of structural parameters which will be determined in our natural history studies.

CONTACTS AND LOCATIONS:
Overall Officials: Chet Whitley, MD, Principal Investigator — University of Minnesota; Michael Mauer, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Universtity of Minnesota, Department of Pediatric Nephrology, Minneapolis, Minnesota